CLINICAL TRIAL: NCT04950231
Title: Investigation on the Knowledge Needs of ALS Patients and Their Caregivers at Home
Brief Title: Investigation on Home Care Needs of ALS Patients and Their Caregivers
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2020082
Record Dates: First submitted 2021-06-27; First posted 2021-07-06 (Actual); Last update posted 2021-07-06 (Actual); Status verified 2021-06

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: The questionnaire survey — Questionnaires were issued and collected by 6 competent nurses with strict training, data entry by 2 researchers, statistical analysis by 1 researcher, and quality control by the other 2 researchers throughout the process.

SUMMARY:
The research target

1. To investigate the home nursing knowledge needs of ALS patients;
2. Investigate the needs of ALS caregivers for home nursing knowledge;
3. To compare the differences between patients and caregivers in the knowledge needs of patients' refusal to care, so as to provide patients and caregivers with targeted care, meet the needs of patients, improve the quality of life of patients, and extend the survival period.

DETAILED DESCRIPTION:
The research target

1. To investigate the home nursing knowledge needs of ALS patients;
2. Investigate the needs of ALS caregivers for home nursing knowledge;
3. To compare the differences between patients and caregivers in the knowledge needs of patients' refusal to care, so as to provide patients and caregivers with targeted care, meet the needs of patients, improve the quality of life of patients, and extend the survival period.

Assessment indicators

1. Scale: Self-designed questionnaire "Questionnaire on the Degree of Home Nursing Knowledge Needs of ALS Patients or Their Families";
2. Amyotrophic lateral sclerosis function rating scale (ALS FRS)

ELIGIBILITY:
Inclusion Criteria:

* confirmed and suspected patients of ALS diagnostic criteria revised by E1 Escorial in 1998;Conscious and stable vital signs;Signing the informed consent;

Exclusion Criteria:

* patients with severe medical diseases, such as severe cardiovascular and cerebrovascular diseases, liver and kidney failure, etc.The existing resources cannot complete the questionnaire to fill in the exclusion of patients, but the caregivers can fill in the questionnaire;

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Six rigorously trained nurses in charge will issue and collect the questionnaire, two researchers will enter the data, one researcher will perform statistical analysis of the data, and the other two researchers will control the quality of the whole process.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Scale | 1 year after recruitment
  Scale: Self-designed questionnaire Questionnaire on the Degree of Home Nursing Knowledge Needs of ALS Patients or Their Family Members;

SECONDARY OUTCOMES:
(ALS FRS) | 1 year after recruitment
  Amyotrophic Lateral Sclerosis Function Scale (ALS FRS)

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Yniversity Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No